CLINICAL TRIAL: NCT05417256
Title: A Prospective Randomized Trial Comparing the Application of Arndt and Tappa Endobronchial Blocker During Pediatric One Lung Ventilation
Brief Title: Comparing Arndt and Tappa Endobronchial Blocker During Pediatric One Lung Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Meltem Savran Karadeniz, Associated Professor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/930
Record Dates: First submitted 2022-06-05; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Lung Diseases
Keywords: Arndt endobronchial blocker; Tappa endobronchial blocker; Pediatrics; One lung ventilation; Thoracic Surgery
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tappa Blocker Group (Active Comparator): After orotracheal intubation, Tappa endobronchial blocker will be inserted using a broncoscope by an experienced anaesthetist. Time from laryngoscopy to successful placement of the endobronchial blocker will be recorded.
  Interventions: Device: Tappa Endobronchial Blocker
- Arndt Blocker Group (Active Comparator): After orotracheal intubation, Arndt endobronchial blocker will be inserted using a broncoscope by the experienced anaesthetist. Time from laryngoscopy to successful placement of the endobronchial blocker will be recorded.
  Interventions: Device: Arndt Endobronchial Blocker

INTERVENTIONS:
Device: Tappa Endobronchial Blocker — After intubation, the Tappa bronchial blocker will be advanced either through the intubation tube or outside the tube using a fiberoptic broncoscope. Once the position of the blocker is confirmed, the cuff of the blocker will be inflated with 1-3 mL of air. Since Tappa blocker has an autoinflation system, the anaesthetist can both inflate the cuff with one hand and operate the fiberoptic broncoscope at the same time.
  Arms: Tappa Blocker Group
Device: Arndt Endobronchial Blocker — After intubation, the endobronchial blocker will be passed through a multiport airway adapter that is placed at the proximal end of the tracheal tube.The fiberoptic broncoscope will be passed through the port and then through the guidewire loop at the end of the blocker. The bronchial blocker and the broncoscope will be advanced as a single unit into the target part of a right or left lung. The broncoscope will be withdrawn into the trachea and the blocker cuff will be inflated and the position of the blocker will be confirmed using the fiberoptic broncoscope. The wire loop will be removed after correct placement of the blocker. Once the guide wire is removed, the blocker can't be replaced.
  Arms: Arndt Blocker Group

SUMMARY:
This study aims to evaluate the efficacy and ease of placement of two different endobronchial blockers(Arndt and Tappa blocker) for pediatric patients undergoing thoracotomy. Time from laryngoscopy to successful insertion of the blocker by an experienced anaesthetist will be recorded and the difficulty of placement of the blocker will be assesed. We plan to evaluate the lung collapse and also observe the effect of two different bronchial blockers on patients' ventilation and oxygenation and adverse events such as desaturation, failed one lung ventilation.Our primary outcome is the time from laryngoscopy to successful insertion of the bronchial blocker by an experienced anaesthetist. Our secondary outcomes are effects of two different bronchial blockers on lung isolation score, ease of placement of the bronchial blocker, mechanical ventilation parameters (tidal volume, respiratory rate, peak airway pressure, plateau pressure, compliance), intraoperative blood gas analysis (paO2, pCO2, saO2, lac), frequency of malposition after successful blocker placement, surgical exposure and complications.

DETAILED DESCRIPTION:
Many techniques for one lung ventilation exist including the use of double-lumen tubes, endotracheal tubes and bronchial blockers. The choice of lung isolation technique depends on the age, the size of the patient, experience of the anaesthetist and type of the surgery. The use of double lumen tube for one lung ventilation is very common. However, it may be challenging and hazardous in some cases such as pediatric patients, patients with tracheostomy, difficult airway scenarios. Endobronchial blockers can be used for these cases. Bronchial blockers have high-volume,low-pressure balloons so they are less likely to cause damage to the airway mucosa while achieving a successful lung isolation. Arndt blocker has a low-pressure, high-volume balloon, a multiport airway adapter and a guide loop. On the other hand, Tappa bronchial blocker has an auto inflation balloon, and a high volume low pressure cuff. It also has 'Tappa angle' which is designed as per human anatomy which makes it easier to insert.

In our study, we aim to compare the efficacy and ease of placement of Arndt and Tappa blocker for pediatric one lung ventilation. Our primary outcome is the time from laryngoscopy to successful insertion of the bronchial blocker by an experienced anaesthetist. Secondary outcomes are effects of two different bronchial blockers on lung isolation score, ease of placement of the bronchial blocker, mechanical ventilation parameters (tidal volume, respiratory rate, peak airway pressure, plateau pressure, compliance), intraoperative blood gas analysis (paO2, pCO2, saO2, lac), frequency of malposition after successful blocker placement, surgical exposure and complications. The difficulty of placement of the blocker will be assesed by a 5-point scale (1:very easy, 5:impossible) and the lung collapse will be evaluated by using a 10-point scale (10: complete collapse).

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing thoracic surgery
* American Society of Anesthesiology Class 1-2-3

Exclusion Criteria:

* Denial of patients or parents
* Coagulopathy
* With preexisting cardiac dysfunction
* Wtih history of renal and/or hepatic dysfunction

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-07-25 (Estimated); Primary Completion 2022-12-25 (Estimated); Study Completion 2023-10-20 (Estimated)

PRIMARY OUTCOMES:
Time from laryngoscopy to placement of the bronchial blocker | Up to 30 minutes
  Time from laryngoscopy to correct insertion of the bronchial blocker by an experienced anaesthetist will be recorded.

SECONDARY OUTCOMES:
Lung collapse score | Up to 30 minutes
  Lung collapse will be assesed at 5,10,15,and 20 minutes after pleural opening using a 10-point scale by the surgeon. 1 point refers to the inflated lung and 10 point refers to a completely collapsed lung.
Difficulty of placement | Up to 30 minutes
  The anaesthetist will rate the difficulty of placement of the bronchial blocker using a 5-point scale, 1 point being very easy and 5 points being impossible to insert.
Tidal volume | Up to 120 minutes
  Volume of gas delivered during each ventilator breath.
Respiratory rate | Up to 120 minutes
  Number of breaths delivered by the ventilator per minute.
Peak airway pressure | Up to 120 minutes
  Pressure used to deliver tidal volume by overcoming resistance in airways and lungs .
Plateau pressure | Up to 120 minutes
  End inspiratory pressure during a period with no gas flow in the circuit.
Compliance | Up to 120 minutes
  Change in volume of the lung produced by a change in pressure across the lung.
Partial pressure of oxygen | At 15 minutes after initiation of one lung ventilation.
  Measurement of oxygen pressure in arterial blood.
Partial pressure of carbon dioxide | At 15 minutes after initiation of one lung ventilation.
  Measurement of carbon dioxide pressure in arterial blood.
Lactate | At 15 minutes after initiation of one lung ventilation.
  Lactate levels in arterial blood gas is used to evaluate tissue perfusion.
Frequency of malposition of the bronchial blocker | Up to the end of one lung ventilation intraoperatively.
  Frequency of malposition of the bronchial blocker after successful bronchial blocker placement will be recorded if the blocker displaces.
Length of intensive care unit (ICU) stay | Up to 48 hours
  If the patients stay in ICU postoperatively
First mobilitisition time | Up to 24 hours
  First mobilitisition time
Length of hospital stay | Up to 1 week
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Savran Karadeniz, Assoc Prof, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Baek SY, Kim JH, Kim G, Choi JH, Jeong CY, Ryu KH, Park DH. Successful one-lung ventilation by blocking the right intermediate bronchus in a 7-year-old child: a case report. J Int Med Res. 2019 Jun;47(6):2740-2745. doi: 10.1177/0300060519845782. Epub 2019 May 8. PMID 31068034
- [Result] Wu C, Liang X, Liu B. Selective pulmonary lobe isolation with Arndt pediatric endobronchial blocker for an infant: A case report. Medicine (Baltimore). 2019 Dec;98(50):e18262. doi: 10.1097/MD.0000000000018262. PMID 31852095
- [Result] Fabila TS, Menghraj SJ. One lung ventilation strategies for infants and children undergoing video assisted thoracoscopic surgery. Indian J Anaesth. 2013 Jul;57(4):339-44. doi: 10.4103/0019-5049.118539. PMID 24163446
- [Result] Cay DL, Csenderits LE, Lines V, Lomaz JG, Overton JH. Selective bronchial blocking in children. Anaesth Intensive Care. 1975 May;3(2):127-30. doi: 10.1177/0310057X7500300208. PMID 1155755
- [Result] Wald SH, Mahajan A, Kaplan MB, Atkinson JB. Experience with the Arndt paediatric bronchial blocker. Br J Anaesth. 2005 Jan;94(1):92-4. doi: 10.1093/bja/aeh292. Epub 2004 Oct 14. PMID 15486004
- See also: Selective pulmonary lobe isolation with Arndt pediatric endobronchial blocker for an infant — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC6922580/
- See also: One lung ventilation strategies for infants and children undergoing video assisted thoracoscopic surgery — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3800324/
- See also: Selective bronchial blocking in children — http://pubmed.ncbi.nlm.nih.gov/1155755/
- See also: Experience with the Arndt paediatric bronchial blocker — http://pubmed.ncbi.nlm.nih.gov/15486004/
- See also: Successful one-lung ventilation by blocking the right intermediate bronchus in a 7-year-old child: a case report — http://pubmed.ncbi.nlm.nih.gov/31068034/